CLINICAL TRIAL: NCT00545922
Title: Cognitive Behavior Therapy for Anxiety and Depression for Patients With Chronic Obstructive Pulmonary Disease (COPD): A Randomized, Controlled Clinical Trial in an Outpatient Pulmonary Clinic.
Brief Title: Cognitive Behavioral Therapy for Anxiety and Depression in COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bergen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REK 3.2007.1668
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-10

CONDITIONS: Anxiety; Depression; Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; anxiety; depression; cognitive behavioral therapy
MeSH Terms: conditions — Anxiety Disorders; Depression; Pulmonary Disease, Chronic Obstructive | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 7 weekly sessions of group cognitive behavioral therapy
  Interventions: Behavioral: Cognitive behavioral therapy
- B (Active Comparator): Minimal Telephone Contact
  Interventions: Behavioral: Minimal Telephone Contact

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Seven weekly sessions (2 hrs) in groups
  Arms: A
Behavioral: Minimal Telephone Contact — Telephone contact (max. 10 minutes) every other week during the 7-week intervention
  Arms: B

SUMMARY:
The purpose of this study was to examine the efficacy of manualized, short-term group cognitive behavioral therapy for COPD patients suffering from clinically significant symptoms of anxiety and/or depression.

DETAILED DESCRIPTION:
Anxiety and depressive disorders have been demonstrated in 16-50% of patients with chronic obstructive pulmonary disease (COPD), and clinically significant levels of anxiety or depressive symptoms seem to be even more common.Despite the multiple, severe consequences, majority of COPD patients with co-morbid anxiety or depression do not seem to receive any treatment for the psychological disturbance.

Cognitive behavioral therapy (CBT) is a well-known approach for treating anxiety and depression, and data has demonstrated effectiveness of CBT for older individuals with anxiety. CBT has also improved exercise tolerance compliance in COPD patients, and pilot studies using CBT components have shown effectiveness in improving mental health and functional status for patients with COPD.

Given the increasing number of patients suffering from COPD and the high prevalence of anxiety and depression in the population, the current study was designed to examine the efficacy of CBT in groups for anxiety and depression in patients with COPD. At present, CBT-based interventions focusing on mental health symptoms are not widely available for COPD patients, and the potential of CBT for improving emotional well-being is not systematically considered in existing treatment alternatives. The study expands the findings from previous pilot studies by focusing on COPD patients with clinically significant levels of anxiety and depression. The wide breadth of coping skills included in the CBT intervention target symptoms of both anxiety and depression, and thus the utility of the intervention for managing mental health symptoms is not restricted to any specific DSM-IV diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* 40 years or older
* scores of 16 or higher on the Beck Anxiety Inventory and/or 14 or higher on the Beck Depression Inventory II
* COPD diagnosis

Exclusion Criteria:

* participation in other studies likely to influence the patient in terms of confounding effects
* signs of cognitive impairment defined by a score of less than 23 on the Mini-Mental State Examination
* presence of psychotic disorders, non-nicotine substance use disorders, bipolar disorders, or suicidal intentions as identified by clinical assessment based on the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (SCID-I/P)
* having a serious somatic condition preventing active participation in the present study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-04; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory | Intervention period of 8 weeks, 6 month follow-up
Beck Depression Inventory-II | Intervention period of 8 weeks, 6 month follow-up

SECONDARY OUTCOMES:
St. George's Respiratory Questionnaire | Intervention period of 8 weeks, 6 month follow-up
Pittsburgh Sleep Quality Inventory | Intervention period of 8 weeks, 6 month follow-up
Actigraphy (Sleep effectiveness) | Intervention period of 8 weeks, 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Inger Hilde Nordhus, Dr. philos, Study Director — University of Bergen
Locations (1):
- Outpatient pulmonary clinic, Haukeland University Hospital, Bergen, Norway